CLINICAL TRIAL: NCT03903367
Title: Bilateral Continous Thoracic Paravertebral Block Versus IV Fentanyl Infusion For Perioperative Analgesia in Patients Undergoing Cardiac Surgery Through Median Sternotomy
Brief Title: Thoracic Paravertebral Block Versus IV Fentanyl Infusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa Rashwan, Samaa Abou Alkassem Rashwan, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Beni-Suef Hospital
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): standard GA and receive fentanyl infusion 2 mcg/kg/h after tracheal intubation and stopped at the end of the operation ,When HR or MBP increased ≥20% from base line readings, incremental dose of fentanyl will be given (2mcg /kg).
  Interventions: Drug: Fentanyl Citrate
- paravertebral block (Active Comparator): Bilateral thoracic paraverteberal catheters will be inserted preoperative at level of T4 in order to block thoracic dermatomal levels from T3-T7 and 0.3ml/kg 0.25% bupivacaine bouls dose in each catheter maximum 20 ml in each catheter before induction and testing sensation bilaterally by pinprick and ice after 15-20min from injection then standard GA and after tracheal intubation continuous infusion of 0.1 ml /kg/h 0.25% bupivacaine in each catheter and stopped at the end of the operation , When HR or MBP increased ≥20% from base line readings, increamental dose of fentanyl will be given (2mcg /kg), the catheters will be removed after 24 h.
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Fentanyl Citrate — standard GA and receive fentanyl infusion 2 mcg/kg/h after tracheal intubation and stopped at the end of the operation ,When HR or MBP increased ≥20% from base line readings, incremental dose of fentanyl will be given (2mcg /kg).
  Other Names: fentanyl

SUMMARY:
High-quality analgesia during and following cardiac surgery is infrequently obtained, Sternotomy and thoracotomy is associated with significant pain that resulte in hypoventilation, atelectasis, and hypoxemia,Pain management is rarley a priority in the immediate postoperative care of these patients, who frequently require mechanical ventilation in an intensive care environment

DETAILED DESCRIPTION:
Paravertebral nerve blocks (PVBs) can provide excellent intraoperative anaesthetic and postoperative analgesic conditions with less side effects and fewer contraindications than central neural blocks,Bilateral PVB has been successfully used in the thoracic, abdominal, and pelvic regions(12). Paravertebral analgesia is produced by placing local anaesthetic (LA) alongside the vertebral column, close to the exit of the spinal nerves(13)..

Traditionally, profound intraoperative analgesia has been provided by using high doses of opioids to suppress hormonal and metabolic stress responses to surgical stimuli. This regimen resulted in improved morbidity and mortality after cardiac surgery(14).

ELIGIBILITY:
Inclusion Criteria:

* males and females patients scheduled for elective open heart surgery

Exclusion Criteria:

* Patients with chest trauma, injuries to peripheries, unstable hemodynamics, sensitivity to local anesthetic drugs, infection at the operation site, renal or hepatic dysfunction, left ventricular dysfunction, coagulation abnormalities and patients on opioids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Critical-Care Pain Observation Tool | Critical-Care Pain Observation Tool (CPOT) will be assessed 1 hour after admitting the patient to the ICU, as base line reacord then every 4 hoursfor 24 hours
  The aim of this study is to compare the efficacy of continuous bilateral thoracic paravertebral block and IV fentanyl infusion on perioperative pain in patients subjected to conventional cardiac surgery through median sternotomy

CONTACTS AND LOCATIONS:
Overall Officials: Samaa ak Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No